CLINICAL TRIAL: NCT03474666
Title: Postoperative Glycemic Control and the Surgical Site Infection Incidence Among Liver Transplantation Recipients: Randomized Clinical Trial
Brief Title: Glycemic Control and Surgical Site Infection Incidence Among Liver Transplantation Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The data safety monitoring inboard recommended stopping the study.
Sponsor: Ramon Oliveira (Other)
Responsible Party: Sponsor-Investigator, Ramon Oliveira, Ph.D Candidate at University of Sao Paulo School of Nursing, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80351717.7.0000.5392; U1111-1210-2322 (Other: Universal Trial Number - World Health Organization)
Record Dates: First submitted 2018-03-02; First posted 2018-03-22 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Liver Transplantation; Surgical Wound Infection
Keywords: Liver Transplantation; Surgical Wound Infection; Hiperglycemia
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Insulin initially as continuous infusion/subcutaneous for first 24-48 hours followed by subcutaneous administration once subjects eating until hospital discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strict Glycemic Control Group (Active Comparator): Intravenous insulin as described by Keegan and Cols. 2010.
  Interventions: Procedure: Strict Glycemic Control Group
- Standard Glycemic Control Group (Active Comparator): Subcutaneous insulin as instititional protocol.
  Interventions: Procedure: Standard Glycemic Control Group

INTERVENTIONS:
Procedure: Strict Glycemic Control Group — The strict protocol adopted to conduct the study was proposed by Keegan e Cols.(2010) to be used among adult LT recipients that consist of a continuous intravenous insulin infusion. The targeted blood glucose range is 80-130 mg/dL. The procedure must be stopped when the patient can ingest at least 50% of liquid diet or receive bolus tube feedings.
  Arms: Strict Glycemic Control Group
Procedure: Standard Glycemic Control Group — The targeted blood glucose range is 130-180 mg/dL
  * Blood glucose reading: ≤ 180 mg/dL - subcutaneous insulin dose: 0
  * Blood glucose reading: ≥181 mg/dL and ≤250 mg/dL - subcutaneous insulin dose: 5 IU
  * Blood glucose reading: ≥251 mg/dL and ≤300 mg/dL - subcutaneous insulin dose: 10 IU
  * Blood glucose reading: ≥301 - subcutaneous insulin dose: 15 IU
  Arms: Standard Glycemic Control Group

SUMMARY:
Context: The hyperglycemia is an important independent risk factor for the Surgical Site Infection (SSI) development among liver transplantation recipients. Objective: To evaluate the effects of an intensive postoperative protocol of blood glucose management on the surgical site infection incidence among liver transplantation recipients. Material and methods: It is an open-label clinical trial that will be randomized into 2 groups of blood glucose (BG) control: patients will undergo BG control regular in the facility chosen to research development (BG targeted 130-180 mg/dL) and the second one will undergo intensive BG control (BG targeted 80 - 130 mg/dL) until patients are eating at least 50% of a full liquid diet or receiving bolus tube feedings. A computer program will be employed to generate the randomized schedule that will be put into sequentially numbered opaque sealed envelopes by an external expert to research. A finger prick device will be used to measure the blood glucose. A blinded adjudication committee to analyse the primary endpoint SSI will adopt the SSI criteria given by the Centers for Disease Control and Prevention. The research proposal will be registered on ClinicalTrials.gov database. Central tendency and dispersion measures, Pearson's χ2 test, Fisher's Exact Test, Mann-Whitney, Wilcoxon-Mann-Whitney and survival analysis by Kaplan-Meier estimated and Log-rank test will be used for data analyses. Expected outcomes: The results of the study should contribute to establishing better clinical practices on glycemic control in the liver transplantation recipient's postoperative period aiming to reduce SSI incidence and its associated morbidity and mortality.

DETAILED DESCRIPTION:
The Surgical Site Infections (SSI's) are the most frequent healthcare-associated infections and are an important infectious complication in the postoperative period among liver transplantation (LT) recipients. SSI incidence among LT recipients, whose allografts were from deceased donors, varied from 9.6% to 35.5% according to a recent literature review. In general surgical procedures, SSI increases the length of stay, morbidity and healthcare costs. Besides that, among LT recipients SSI can raise the risks of the allografts dysfunctions, acute rejections and as a consequence a reduction in the recipient's survival.

There are several risk factors for SSI among LT recipients. There is a relationship among supply sterilization quality, the characteristics of surgical procedure, the operation room environment as well as the allograft's and recipient's conditions and SSI occurrence. In regard to LT recipients, results from previous research highlighted hyperglycemia as an important independent predictor of SSI. Furthermore, regarding this population, it is known from observational studies that LT recipients affected by hyperglycemia are exposed, approximately, to three times the risk of SSI comparatively to LT recipients not exposed.

The concern about maintaining normoglycaemia in acute care facilities is not recent; several studies have been done including on clinical and surgical patients from some medical specialities showing the morbidity and mortality reduction throughout the adoption of strict glycaemic control protocols.

However, among critical surgical patients the LT recipients are highlighted; since they are exposed to impairment in blood glucose metabolism in the perioperative period as a consequence of an intraoperative acute stress state, blood loss and transfusions, the reperfusion phase, use of glucocorticoids and catecholamines.

Results from previous studies pointed the hyperglycaemia among LT recipient as a frequent complication, 94% of them presented it at least once in the transplantation's postoperative period.

The high blood glucose levels can produce electrolyte and acid-base disturbances besides altered plasmatic distribution of sodium. There are impairments to the white blood cells activities, such as reduction in the adherence, chemotaxis, phagocytosis and superoxide formation. Lymphocytes apoptosis combined with T-cell activities suppression besides attenuation of immunoglobulin's work as a consequence of glycosylation.

In spite of evidence from laboratory studies that indicate remarkable impairments caused by hyperglycemia in immune model animals immunologic system, uncertainties remain to evaluate the glycaemic control as a strategy for SSI prevention. Analysing the guidelines to prevent SSI published by World Health Organization, Centers for Disease Control and Prevention (United States of America), National Institute for Health and Care Excellence (United Kingdom), Society for Healthcare Epidemiology of America (United States of America) and Brazilian Health Regulatory Agency conditional recommendation regard the adoption of strategies to strict glycaemic control in the postoperative phase, besides there is no consensus about how glycaemic level could work as a protective factor for SSI among patients who underwent general surgeries.

Moreover, there have been few investigations evaluating the hyperglycaemia effects or blood glucose control in the postoperative phase of LT recipients. Besides the few studies concerned on the topic among LT recipients, the majority of them were observational studies, designed as retrospective cohorts, which could compromise the body's evidence quality. Also, in the previous studies enrolled patients underwent liver-kidney transplantation, which can cause a negative impact on the effects of glycemic control analyses and there is research where recipients presented lower means of Model for End-Stage Liver Disease (MELD) from 19.0 to 28.2 that are lower MELD means than the observed in Brazilian transplantation centres. Finally, we observed the absence of clear criteria for SSI diagnosis in some studies.

It is known that the preoperative screening in living donor LT of donors and recipients as baseline characteristics are different of LT whose allografts came from deceased donors; for instance, liver-kidney recipients who undergo to distinct immunosuppression schemes. Furthermore, lower MELD scores represent LT recipients that could be exposed to diverse risk factors for SSI when compared to LT recipients who the MELD score is higher.

Thus, it sounds appropriate that research aiming to evaluate the effect of strict blood glucose control on SSI incidence among LT recipients should be made. In addition, nurse-initiated blood glucose control protocols, among critically ill patients, are frequently developed. And, a recent literature review pointed to the lack of prospective studies that addressed the evaluation of the outcomes of strict glycaemic control among LT recipients on SSI incidence.

The study hypothesis is: the postoperative strict glycaemic control reduces the SSI incidence among LT recipients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of LT whose allograft came from deceased donors
* Able to give informed consent personally or via a family member who has appropriate authorization to do so if patient unconscious.
* Blood glucose level over 130 mg/dL in the first 24 hours postoperatively

Exclusion Criteria:

* The patients that underwent any kind of surgery with or without prosthesis implant in the 30 days before the LT
* Recipients submitted to multiple organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | SSI occurs within 30 days after the LT
  Surgical site infection following the Centers for Disease Control and Prevention defining criteria (2018)

SECONDARY OUTCOMES:
Hyperglycemia | During first 48h ICU stay
  Hyperglycemia > 250 mg/dL
Hypoglycemia | During first 48h ICU stay
  Hypoglycemia < 60 mg/dL
Duration of mechanical ventilation | Within 30 days after LT
  Duration of mechanical ventilation through postoperative ICU stay
ICU stay | Within 30 days after LT
  ICU stay until 30 days after LT
Ward stay | Within 30 days after LT
  Postoperative ward stay
Death | 90 days after LT
  Death within 90 days after LT
Surgical Site Infection or death | Surgical site infection within 20 days following liver transplantation or death within 90 days following liver transplantation
  Surgical site infection following the Centers for Disease Control and Prevention defining criteria (2018)
Hospital length of stay | Until 100 weeks after liver transplantation
  Time between the hospital admission to liver transplantation and hospital discharge

OTHER OUTCOMES:
PPI preoperative use and SSI | Preoperative period
  Proton-pump inhibitor and ocurrence of SSI

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa B Poveda, Ph.D, Study Chair; Judith Tanner, Ph.D, Study Director; Jorge M Padilla, M.Sc, Study Director
Locations (1):
- Hospital Santa Casa de São José dos Campos, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira RA, Tanner J, Mancero JMP, de Brito Poveda V. Effects of Intensive Blood Glucose Control on Surgical Site Infection for Liver Transplant Recipients: A Randomized Controlled Trial. Transplant Proc. 2023 Jan-Feb;55(1):170-177. doi: 10.1016/j.transproceed.2022.10.062. Epub 2022 Dec 24. PMID 36567173
- See also: Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017 — http://www.ncbi.nlm.nih.gov/pubmed/28467526
- See also: Effect of antibiotic prophylaxis on the risk of surgical site infection in orthotopic liver transplant — http://www.ncbi.nlm.nih.gov/pubmed/18508358
- See also: The effect of surgical site infections on outcomes and resource utilization after liver transplantation — http://www.ncbi.nlm.nih.gov/pubmed/11490376
- See also: Risk factors for development of surgical site infections among liver transplantation recipients: An integrative literature review — http://www.ncbi.nlm.nih.gov/pubmed/28689978
- See also: Bacteremia and septic shock after solid-organ transplantation. — http://www.ncbi.nlm.nih.gov/pubmed/16386636
- See also: The direct and indirect effects of infection in liver transplantation: pathogenesis, impact, and clinical management. — http://www.ncbi.nlm.nih.gov/pubmed/12520651
- See also: Causes of mortality after liver transplantation: a single center experience in mainland china. — http://www.ncbi.nlm.nih.gov/pubmed/21940379
- See also: Safety and effectiveness of intensive insulin protocol use in post-operative liver transplant recipients. — https://www.ncbi.nlm.nih.gov/pubmed/20832556

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03474666/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03474666/SAP_001.pdf